CLINICAL TRIAL: NCT06577220
Title: A Randomized Controlled Trial of Mailed Self-Sample HPV Testing to Increase Cervical Cancer Screening Participation Among Minority/Underserved Women in an Integrated Safety Net Healthcare System Asian/Asian American Women
Brief Title: Prospective Evaluation of Self-Testing to Increase Screening (PRESTIS) Asian/Asian American Women Supplement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jane Montealegre, Associate Professor, M.D. Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: H-44944 S1
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer; Human Papillomavirus Infection
Keywords: Screening; Human Papillomavirus Infection; Self-Testing
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Telephone Recall (Active Comparator): Participants receive a scripted telephone recall from a trained patient navigator on behalf of Harris Health System
  Interventions: Behavioral: Telephone Recall
- Mailed HPV Self-Sampling Kit (Experimental): Participants receive a scripted telephone recall from a patient navigator on behalf of Harris Health System and receive a mailed HPV self-sampling kit with a prepaid return envelope
  Interventions: Behavioral: Telephone Recall; Behavioral: Mailed HPV Self-Sampling Kit
- Mailed HPV Self-Sampling Kit + Patient Navigation (Experimental): Participants receive a scripted telephone recall and mailed self-sampling kit with a pre-paid return envelope. Within 3-5 days of the kit's mail-out, participants will receive a telephone call from a patient navigator to provide one-on-one education.
  Interventions: Behavioral: Telephone Recall; Behavioral: Mailed HPV Self-Sampling Kit; Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Telephone Recall — Participants receive a scripted telephone recall from a trained patient navigator.
Behavioral: Mailed HPV Self-Sampling Kit — Participants receive a mailed kit that allows them to self-collect a cervical sample in their home and return it to a laboratory for human papillomavirus (HPV) testing.
  Arms: Mailed HPV Self-Sampling Kit; Mailed HPV Self-Sampling Kit + Patient Navigation
Behavioral: Patient Navigation — Participant receives telephone call from patient navigator within 3-5 days of receipt of self-collection kit. Patient navigator provides one-on-one education on cervical cancer screening and self-collection of cervical sample.
  Arms: Mailed HPV Self-Sampling Kit + Patient Navigation

SUMMARY:
Regularly attending for Pap test cervical cancer screening in a clinic is often unfeasible and/or unacceptable to many women and persons with a cervix. This study is a supplement to increase representation of Asian and Asian American women in a pragmatic clinical trial that evaluates if mailing and testing self-sampled kits for high-risk human papillomavirus (HPV) can cost-effectively increase screening participation among underserved minority women in a safety-net health system.

DETAILED DESCRIPTION:
Regularly attending for Pap test cervical cancer screening in a clinic is often unfeasible and/or unacceptable to many women and persons with a cervix. Using mailed self-sampling kits to test for high-risk human papillomavirus (HPV), the virus that causes cervical cancer, may overcome multiple barriers to clinic-based screening. The parent study (NCT03898167) is a randomized controlled trial to compare the effectiveness of three outreach interventions to increase primary screening participation and clinical follow-up among underscreened women a in a safety net health system. The three strategies that will be evaluated are: 1) telephone recall; 2) telephone recall with mailed self-sample HPV testing kits; and 3) telephone recall with mailed self-sample HPV testing kits and patient navigation. A supplemental accrual of Asian/Asian American persons (target n=240) was added to increase representation of this subpopulation in the parent trial.

ELIGIBILITY:
Inclusion Criteria:

* Asian ethnicity reported in the electronic health record
* no history of hysterectomy or cervical cancer
* no Pap test in the past 3.5 years or Pap/HPV co-test in the past 5.5 years
* patient of Harris Health System in Harris County (Houston), Texas
* have at least 2 visits to ambulatory care within Harris Health System in the past 5 years
* be currently enrolled in a healthcare coverage or financial assistance plan accepted by Harris Health System or have been enrolled in a Harris Health coverage plan in the past 12 months

Exclusion Criteria:

* no valid telephone contact information
* unable to communicate in English, Vietnamese or Spanish
* currently pregnant
* history of cervical dysplasia in the past 3.5 years

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 111 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
Primary screening participation | [Time Frame: within 6 months of randomization
  completion and return of a mailed self-sample HPV testing kit that is adequate for testing (i.e., does not produce unsatisfactory results) or attendance for clinic-based screening

SECONDARY OUTCOMES:
Screening tests results | Time Frame: within 6 months of randomization
  Results of HPV test using self-collected samples (positive, negative, or inadequate)
completion of clinical follow-up among women with an abnormal screening test result | Time Frame: within 12 months of screening test result
  Electronic medical record (EMR)-confirmed attendance for colposcopy among participants who had a positive test by clinic-based screening; EMR- confirmed attendance for colposcopy or subsequent clinic-based screening among those who had a positive test by self-sampling

OTHER OUTCOMES:
Detection of cervical precancer | [Time Frame: within 12 months of screening test result]
  Histologically-confirmed cervical intraepithelial neoplasia grade II or greater (CIN2+)
Treatment of cervical precancer | [Time Frame: within 6 months of diagnosis]
  Treatment of histologically-confirmed cervical intraepithelial neoplasia grade II or greater (CIN2+) per American Society for Colposcopy and Cervical Pathology guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Harris Health System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Within one year of study completion.
Access Criteria: Available upon request to Principal Investigator.

REFERENCES:
- [Background] Montealegre JR, Anderson ML, Hilsenbeck SG, Chiao EY, Cantor SB, Parker SL, Daheri M, Bulsara S, Escobar B, Deshmukh AA, Jibaja-Weiss ML, Zare M, Scheurer ME. Mailed self-sample HPV testing kits to improve cervical cancer screening in a safety net health system: protocol for a hybrid effectiveness-implementation randomized controlled trial. Trials. 2020 Oct 21;21(1):872. doi: 10.1186/s13063-020-04790-5. PMID 33087164